CLINICAL TRIAL: NCT03812809
Title: A Phase IIb, Open-label, Single-arm Study to Assess the Safety and Efficacy of BPI-7711 Capsule in Patients With Metastatic or Recurrent Non-small Cell Lung Cancer With EGFR Mutation and T790M Mutation Positive.
Brief Title: A Phase IIb Study of BPI-7711 Capsule in Non-small Cell Lung Cancer Patients With T790M Mutation Positive
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beta Pharma Shanghai (Industry)
Responsible Party: Sponsor
Organization: Beta Pharma, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPI-7711201
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: NSCLC
Keywords: EGFR; T790M; NSCLC
MeSH Terms: interventions — rezivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPI-7711 (Experimental): BPI-7711: 180mg, QD, oral
  Interventions: Drug: BPI-7711

INTERVENTIONS:
Drug: BPI-7711 — BPI-7711: 180mg, QD, oral
  Other Names: BPI-7711 capsule

SUMMARY:
A phase IIb, open-label, single-arm study to assess the safety and efficacy of BPI-7711 capsule in patients with metastatic or recurrent non-small cell lung cancer with EGFR mutation and T790M mutation positive.

DETAILED DESCRIPTION:
This is a phase IIb, open-label, single arm study assessing the safety and efficacy of BPI-7711 (180 mg, orally, once daily) in China with a confirmed diagnosis of EGFR sensitizing mutation positive and T790M mutation+ unresectable, locally advanced or metastatic NSCLC, who have progressed on prior EGFR-TKIs treatment. The primary objective of the study is to assess the efficacy of BPI-7711 by assessment of ORR according to RECIST 1.1 by an Independent Central Review.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years.
* Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy.
* Radiological documentation of disease progression after the most recent EGFR-TKI treatment administered. Radiological documentation of disease progression after the most recent treatment, or intolerant to current chemotherapy, or unwilling to accept the current treatment.
* At least one non-brain measurable lesion, not previously irradiated that can be accurately measured at baseline. If only one measurable lesion, the baseline CT should be performed before the biopsy or at least 14 days after the biopsy. Prior irradiated lesion can only be used as biopsy lesion after significant progression.
* Documented EGFR mutation (at any time since the initial diagnosis of NSCLC) known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).
* Patients must have central confirmation of tumor T790M mutation+ status from a biopsy sample or a plasma sample taken after confirmation of disease progression on the most recent EGFR-TKI treatment. Primary T790M mutation positive patients should provide prior written evidence before ICF signature and have not received any EGFR-TKI.
* ECOG performance status 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* Females of child-bearing potential using contraception and must have a negative pregnancy test.

Exclusion Criteria:

* Confirmed EGFR 20 exon insertion mutation after the initial diagnosis of NSCLC.
* Treatment with any 1st or 2nd EGFR-TKI (eg, erlotinib, gefitinib, icotinib, afatinib or dacomitinib) within 5x half-life of study entry.
* Treatment with any 3rd generation EGFR TKIs target on T790M mutation.
* Treatment with any cytotoxic chemotherapy, investigational agents, CYP3A4/CYP2C19 potent inhibitor/inducer, or other anticancer drugs within 14 days of study entry.
* Prior medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to study treatment.
* Major surgery within 4 weeks of study entry; radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of study entry.
* Refractory nausea and vomiting, chronic gastrointestinal diseases or bowel resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
ORR according to RECIST 1.1 by an Independent Central Review (ICR) | up to 52 weeks
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by MRI or CT. ORR is the percentage of patients with at least 1 visit response of CR or PR (according to independent review) that was confirmed at least 4 weeks later, prior to progression or further anti-cancer therapy.

SECONDARY OUTCOMES:
ORR according to RECIST 1.1 by investigators | up to 52 weeks
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by MRI or CT. ORR is the percentage of patients with at least 1 visit response of CR or PR (according to independent review) that was confirmed at least 4 weeks later, prior to progression or further anti-cancer therapy.
Disease control rate (DCR) according to RECIST 1.1 | up to 104 weeks
  DCR is the percentage of patients with best response of CR, PR or SD (according to independent review), prior to progression (PD) or further anti-cancer therapy.
Progression free survival(PFS) according to RECIST 1.1 | up to 104 weeks
  PFS is the time from date of first dose until the date of PD (by independent review) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from BPI-7711 therapy or received another anti-cancer therapy prior to progression. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Linyi Cancer Hospital, Linyi, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang S, Wu S, Zhao Y, Chen G, Zhu B, Li X, Wang K, Shi J, Cang S, Yao W, Fan Y, Fang J, Zhang L, Zhou J, Wu L, Zheng R, Huang M, Pan Y, Yang Z, Sun M, Yu H, Wang D, Huang J, Wang L, Shu Y, Chen Z, Liu C, Li J, Liu J, Sun S, Guo Y, Meng Z, Liu Z, Han Z, Wu G, Lu H, Ma R, Hu S, Zhao G, Zhang L, Liu Z, Xie C, Zhong D, Zhao H, Bi M, Yi S, Guo S, Yi T, Li W, Lin Y, Chen Z, Zhuang Z, Guo Z, Greco M, Wang T, Zhou A, Shi Y. Central nervous system efficacy of rezivertinib (BPI-7711) in advanced NSCLC patients with EGFR T790M mutation: A pooled analysis of two clinical studies. Lung Cancer. 2023 Jun;180:107194. doi: 10.1016/j.lungcan.2023.107194. Epub 2023 Apr 17. PMID 37163774
- [Derived] Shi Y, Wu S, Wang K, Cang S, Yao W, Fan Y, Wu L, Huang M, Li X, Pan Y, Yang Z, Zhu B, Chen G, Shi J, Sun M, Fang J, Wang L, Chen Z, Liu C, Li J, Liu J, Sun S, Zhao Y, Guo Y, Meng Z, Liu Z, Han Z, Lu H, Ma R, Hu S, Zhao G, Liu Z, Xie C, Zhong D, Zhao H, Yu H, Zhang L, Bi M, Yi S, Guo S, Yi T, Li W, Lin Y, Shu Y, Chen Z, Guo Z, Greco M, Wang T, Shen H. Efficacy and Safety of Rezivertinib (BPI-7711) in Patients With Locally Advanced or Metastatic/Recurrent EGFR T790M-Mutated NSCLC: A Phase 2b Study. J Thorac Oncol. 2022 Nov;17(11):1306-1317. doi: 10.1016/j.jtho.2022.08.015. Epub 2022 Aug 29. PMID 36049654